CLINICAL TRIAL: NCT00522275
Title: An Open-label Extension Trial to Determine Safety and Efficacy of Long-term Oral SPM 927 in Patients With Partial Seizures
Brief Title: Determine Safety and Efficacy of Long-term Oral Lacosamide in Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0756; 2014-004398-18 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Results first posted 2010-11-22 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2017-07

CONDITIONS: Partial Epilepsies
Keywords: Adjunctive treatment in epilepsy; add-on treatment for epilepsy; partial seizures; AEDs; antiepileptic drugs; seizures
MeSH Terms: conditions — Epilepsies, Partial; Seizures | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Up to 800 mg/day lacosamide (flexible dosing)
  Interventions: Drug: lacosamide

INTERVENTIONS:
Drug: lacosamide — 50mg or 100 mg tablets, up to 800 mg/day given twice daily (BID) throughout the trial

SUMMARY:
The purpose of this trial is to determine whether lacosamide is safe and effective for long-term use in patients with partial-seizures from epilepsy

ELIGIBILITY:
Inclusion Criteria:

* Completion of parent clinical trial for treatment of partial seizures

Exclusion Criteria:

* Receiving any study drug or experimental device other than lacosamide
* Meets withdrawal criteria for parent trial or experiencing ongoing serious adverse event

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2004-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (60):
- United States (60):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - San Francisco, California
  - Englewood, Colorado
  - Fairfield, Connecticut
  - Bradenton, Florida
  - Jacksonville, Florida
  - Maitland, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Golden Valley, Minnesota
  - Saint Cloud, Minnesota
  - Saint Paul, Minnesota
  - Chesterfield, Missouri
  - Somerset, New Jersey
  - Albuquerque, New Mexico
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Beaufort, South Carolina
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Marshfield, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Husain A, Chung S, Faught E, Isojarvi J, McShea C, Doty P. Long-term safety and efficacy in patients with uncontrolled partial-onset seizures treated with adjunctive lacosamide: results from a Phase III open-label extension trial. Epilepsia. 2012 Mar;53(3):521-8. doi: 10.1111/j.1528-1167.2012.03407.x. PMID 22372628
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lacosamide
Started | 308
Completed | 138
Not Completed | 170
Not completed — Adverse Event | 35
Not completed — Lack of Efficacy | 80
Not completed — Subject withdrew consent | 16
Not completed — Protocol deviation | 1
Not completed — Unsatisfactory compliance | 11
Not completed — Lost to Follow-up | 8
Not completed — Other: Subject wants to become pregnant | 2
Not completed — Other: Subject is pregnant | 2
Not completed — Other: Subject relocated | 2
Not completed — Other: Subject arrested | 1
Not completed — Other: Site / clinic closed | 4
Not completed — Other: Travel to / from site difficulty | 3
Not completed — Other: Sponsor request | 2
Not completed — Other: Subject ran out of medication | 1
Not completed — Other: Subject had surgery for epilepsy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lacosamide
Number analyzed (Participants) | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 295
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 162
Region of Enrollment [Number; unit: participants]
  United States | 308

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least 1 Treatment-Emergent Adverse Event (TEAE) During the Treatment Period (Maximum 6 Years)
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: During the Treatment Period (Maximum 6 years)
Population: Of the 308 subjects who entered the study, 308 are included in this summary based on the Safety Set (SS). SS population: number of subjects treated.
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 308
subjects | 288

2. Primary Outcome: Number of Subjects Prematurely Discontinuing Due to a Treatment-Emergent Adverse Event (TEAE) During the Treatment Period (Maximum 6 Years)
Description: as for outcome 1
Time Frame: During the Treatment Period (Maximum 6 years)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 308
subjects | 33

3. Primary Outcome: Number of Subjects Reporting at Least 1 Serious Adverse Event (SAE) During the Treatment Period (Maximum 6 Years)
Description: Serious adverse events are any untoward serious medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: During the Treatment Period (Maximum 6 years)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 308
subjects | 71

4. Secondary Outcome: Median Percentage Change From Baseline in 28-day Seizure Frequency During the Treatment Period (Maximum 6 Years)
Description: Negative changes from Baseline indicate an improvement (i.e., a reduction) in 28-day seizure frequency.
Time Frame: Baseline (8-week Baseline Period from the parent study SP0754 [NCT00136019]), Treatment Period (Maximum 6 years)
Population: Of the 308 subjects who were enrolled/treated in the study, 307 are included in this summary based on the Full Analysis Set (FAS). FAS population: number of subjects treated with at least 1 post-baseline seizure diary day with available data during the SP756 study.
Measure: Median (Full Range); unit: percentage change
Arm/Group | Lacosamide
Number analyzed (Participants) | 307
percentage change | -48.5 [-100.0 to 567.7]

5. Secondary Outcome: Percentage of at Least 50 % Responders During the Treatment Period (Maximum 6 Years)
Description: At least 50 percent response is based on the percentage reduction in 28-day seizure frequency during the Treatment Period of the open-label extension relative to the Baseline Phase of the prior study.
Time Frame: Treatment Period (Maximum 6 years)
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 307
percentage of subjects | 48.2

ADVERSE EVENTS:
Time Frame: Maximum of 6 years
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 71/308
Other Adverse Events (participants affected / at risk) | 265/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=308)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 5 (6)
Asthenia (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Chronic hepatitis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Cystitis (Infections and infestations) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Salpingitis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 11 (13)
Dizziness (Nervous system disorders) | 4 (4)
Status epilepticus (Nervous system disorders) | 3 (3)
Coordination abnormal (Nervous system disorders) | 2 (2)
Complex partial seizures (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (2)
Aggression (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Sleep attacks (Psychiatric disorders) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Priapism (Reproductive system and breast disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 (1)
Vagal nerve stimulator implantation (Surgical and medical procedures) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Gastrooesophagitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=308)
Diplopia (Eye disorders) | 46 (72)
Vision blurred (Eye disorders) | 28 (39)
Nausea (Gastrointestinal disorders) | 56 (78)
Vomiting (Gastrointestinal disorders) | 47 (66)
Diarrhoea (Gastrointestinal disorders) | 25 (32)
Constipation (Gastrointestinal disorders) | 22 (22)
Fatigue (General disorders) | 36 (45)
Irritability (General disorders) | 19 (21)
Gait disturbance (General disorders) | 18 (22)
Nasopharyngitis (Infections and infestations) | 53 (83)
Upper respiratory tract infection (Infections and infestations) | 40 (54)
Sinusitis (Infections and infestations) | 32 (46)
Influenza (Infections and infestations) | 26 (28)
Urinary tract infection (Infections and infestations) | 25 (37)
Bronchitis (Infections and infestations) | 17 (23)
Contusion (Injury, poisoning and procedural complications) | 57 (90)
Fall (Injury, poisoning and procedural complications) | 47 (93)
Skin laceration (Injury, poisoning and procedural complications) | 38 (69)
Joint sprain (Injury, poisoning and procedural complications) | 19 (20)
Excoriation (Injury, poisoning and procedural complications) | 18 (38)
Head injury (Injury, poisoning and procedural complications) | 17 (21)
Weight increased (Investigations) | 17 (17)
Gamma-glutamyltransferase increased (Investigations) | 17 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (46)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (26)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (24)
Dizziness (Nervous system disorders) | 154 (260)
Headache (Nervous system disorders) | 67 (91)
Convulsion (Nervous system disorders) | 44 (62)
Tremor (Nervous system disorders) | 41 (57)
Balance disorder (Nervous system disorders) | 41 (51)
Nystagmus (Nervous system disorders) | 34 (37)
Coordination abnormal (Nervous system disorders) | 26 (30)
Somnolence (Nervous system disorders) | 25 (28)
Memory impairment (Nervous system disorders) | 20 (21)
Depression (Psychiatric disorders) | 35 (45)
Insomnia (Psychiatric disorders) | 28 (38)
Anxiety (Psychiatric disorders) | 17 (20)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 (29)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (23)
Rash (Skin and subcutaneous tissue disorders) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.